CLINICAL TRIAL: NCT03371953
Title: Efficacy of Atracurium-vecuronium Combination in Patients Undergoing Laparoscopic Surgery:a Randomised Controlled Study
Brief Title: Evaluation of Atracurium-vecuronium Combination in Laparosocpic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Amitabh Dutta, Senior Consultant & Professor, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EC/10/17/1280
Record Dates: First submitted 2017-12-02; First posted 2017-12-13 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Patients Undergoing Laparoscopic Surgery
Keywords: vecuronium; atracurium; combination
MeSH Terms: interventions — Vecuronium Bromide; Atracurium

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into three groups in a 1:1:1 distribution undertaken by a computer-generated random number system.
  Vecuronium group - 0.08mg/kg vecuronium alone
  Atracurium group- 0.6mg/kg atracurium alone
  Vecuronium-atracurium group- 0.04mg/kg vecuronium and 0.3 mg/kg atracurium combination
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient, the attending anaesthesiologist, and the personnel recording the assessment parameters will be blinded to the randomisation sequence and the drug inside the 5-ml solution is supplied in a 5-ml syringe. The study drug for the three group allocation will be contained in a similar 5-ml solution (drug+0.9% saline solution).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vecuronium group (Active Comparator): Vecuronium 0.08 mg/kg will be administered at induction of anaesthesia for facilitating muscle relaxation
  Interventions: Drug: Vecuronium
- Atracurium group (Active Comparator): Atracurium 0.6 mg/kg will be administered at induction of anaesthesia for facilitating muscle relaxation
  Interventions: Drug: Atracurium
- Vecuronium-Atracurium group (Active Comparator): Vecuronium 0.04 mg/kg + atracurium 0.3 mg/kg will be administered at induction of anaesthesia for facilitating muscle relaxation
  Interventions: Drug: Vecuronium + Atracurium

INTERVENTIONS:
Drug: Vecuronium — A top-up dose of vecuronium will be administered when the TOF count is 1 on the accelerometer. However, if there is a diaphragmatic contraction which interferes with surgical procedure then a dose will be given irrespective of the TOF count.
  Arms: Vecuronium group
Drug: Atracurium — A top-up dose of vecuronium will be administered when the TOF count is 1 on the accelerometer. However, if there is a diaphragmatic contraction which interferes with surgical procedure then a dose will be given irrespective of the TOF count.
  Arms: Atracurium group
Drug: Vecuronium + Atracurium — A top-up dose of vecuronium + atracurium will be administered when the TOF count is 1 on the accelerometer. However, if there is a diaphragmatic contraction which interferes with surgical procedure then a dose will be given irrespective of the TOF count.
  Arms: Vecuronium-Atracurium group

SUMMARY:
Non-depolarising muscle relaxants are routinely employed to provide skeletal muscle relaxation during general anaesthesia (GA). Generally investigators use one or the other type of relaxant agent for this purpose and they are categorised based on their duration-of-action. Atracurium and vecuronium are two common muscle relaxant used during GA. They have an intermediate duration of action (around 40 minutes). Though they are effective relaxants and easy to reverse with reversal agents after the surgery, in case of the common laparoscopy procedures lasting an hour, they are relatively inefficient. There is evidence that when these agents are combined together (in 1:1 ratio), the duration-of-action, and reversibility improves. To render atracurium and vecuronium more efficient with laparoscopic surgery, the proposed study is aimed to evaluate the effects of combining 1/2 the respective standard doses of atracurium and vecuronium given together, in terms of its effect on the onset of block, duration-of-action, and reversibility of the neuromuscular blockade in adults undergoing laparoscopic surgery under GA. The study will be conducted with objective assessment parameter evaluation by TOF Watch SX (Organon, Teknica BV, Boxtel, The Netherlands), which will be used for facilitating institution, control, and monitoring the neuromuscular blockade during surgery. The objective of this study is to evaluate the additive effect of atracurium-vecuronium combination and profile its impact in patients undergoing laparoscopic surgery, especially in terms of increase in duration-of-action of muscle relaxation with the combination of drugs, when compared to respective individual drugs.

DETAILED DESCRIPTION:
The principal pharmacological effect of neuromuscular blocking drugs is to interrupt the transmission of nerve impulses at the neuromuscular junction. They are classified into depolarising (mimics the action of acetylcholine) and non-depolarising (interfere with the action of acetylcholine).In general, we use vecuronium (0.08mg/kg) or atracurium (0.5mg/kg), which are intermediate-acting non-depolarising neuromuscular blocking agents for skeletal muscle relaxation.

The main use of neuromuscular blocking drugs is to provide skeletal muscle relaxation for facilitation of intubation of the trachea and to improve surgical working conditions in the anaesthetised patients. A 2×ED95 dose of non-depolarising muscle relaxant is recommended to facilitate tracheal intubation. In practice, 90% suppression of the single twitch response is usually considered clinical evidence of adequate drug-induced skeletal muscle relaxation.

Laparoscopy has become the most preferred means of surgical access for a variety of procedures. There are many laparoscopic surgeries that last about an hour. But the duration-of-action of bolus (intubating) dose of atracurium or vecuronium when used alone is not sufficient to last for an hour. As a result, for surgeries lasting an hour(e.g. laparoscopic cholecystectomy, laparoscopic total extra-peritoneal repair, etc.), one either end up giving a top up (maintenance) dose of vecuronium/atracurium to extend muscle relaxation or withhold the add-on dose and continue with surgery towards completion. While in the former situation, the anaesthesiologist is required to wait for long even though the surgery is completed; in the latter, either the surgery gets disturbed due to patient's movement (e.g. coughing, bucking) or there may be associated hemodynamic activation, which requires deepening of anaesthesia plane; both harbinger for patient-related adversity.

There are studies which have evaluated the effect of combining two non-depolarizing neuromuscular relaxants on the profile of skeletal muscle relaxation pertinent to anaesthetic (tracheal intubation) and surgical conditions.Atracurium and vecuronium are the most common non- depolarizing muscle relaxants we routinely employ during general anaesthesia (GA). Till date, to our knowledge, there are a very few studies that have evaluated combination of atracurium and vecuronium given together.Though, the limited number of studies which analysed effects of combined neuromuscular relaxation with atracurium and vecuronium underlined that there is an additive effect, commented only on onset-of-action and reversibility of muscle relaxation effect. In addition, no study has yet evaluated the duration-of-action of atracurium- vecuronium combination in adults undergoing laparoscopic surgeries. Muscle relaxation is used for optimising laparoscopic operating conditions by preventing diaphragmatic movement due to irritation by the presence of pneumoperitoneum and achieving more intra-abdominal space for a particular intra-abdominal insufflation pressure. In this context, deeper than normally maintained level of neuromuscular blockade appears to be superior. The investigators contend that combining vecuronium and atracurium would not only facilitate increase in duration-of-action of the relaxation but also provide quality muscle relaxation for the duration of surgery.

The proposed study looks forward to analyse the effect of muscle relaxation profile of vecuronium-atracurium combination versus vecuronium-alone or atracurium-alone in patients undergoing laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I and II
2. Laparoscopic surgeries likely to last for 1 hour duration

Exclusion Criteria:

1. Patient refusal
2. ASA physical status III and IV
3. History of hypersensitivity to atracurium or vecuronium
4. Alcoholism and drug addiction
5. Neuromuscular disorders
6. Neuropsychiatric patients
7. Hepatic and renal disease patients
8. Obese patients
9. Abnormal airway anatomy
10. Risk of oesophageal reflux

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-12-20 (Estimated); Primary Completion 2018-10-25 (Estimated); Study Completion 2018-10-25 (Estimated)

PRIMARY OUTCOMES:
Duration-of-action of the intubating dose | From the time of administration of (0-hours, baseline) till 60-minutes intraoperatively
  Duration of action will be calculated from the time the drug is administered till theTOF count is 1 on the accelerometer.

SECONDARY OUTCOMES:
Onset-of-action of muscle relaxation following intubating dose | From the time of administration of (0-hours, baseline) till 5-minutes intraoperatively
  Onset-of-action will be calculated from the time the drug is administered till theTOF count is 0 on the accelerometer.
Qualitative intubating conditions. | From the time of administration of (0-hours, baseline) till 5-minutes intraoperatively
  Quality of intubating condition will be assessed using 3-point modified Cooper's scale. The intubating conditions will be graded as excellent, good & poor.
  1. The scale "Intubating conditions following intubating dose of non-depolarizing muscle relaxant" is modified from Cooper's Scale. The scale's name is derived from the name of the investigator (Cooper R) who first used it. (Br J Anaesth 1992; 69: 269-73)
  2. The Cooper Scale includes five major variable sets [1. Laryngoscopy (Jaw Relaxation), 2.Vocal-cord position, 3. Vocal cord movement, 4. Reaction to intubation and/or cuff inflation 5. Movement of limbs/ coughing] which are classified as poor, good or excellent. For ease of the study analysis, poor is scored '0', good is scored '1', and excellent is scored '2'. Therefore, each variable has subscale range of 0-2 and, five variables are together ranged as 0-10.
  3. Each of the five subscale range, i. e. 0-2, are added up to gain a 'total scale range score' of 0-10.
Reversibility of muscle relaxant effect | From the time of administration of (0-hours, baseline) till 5-minutes post administration
  Time for complete reversal of effect of muscle relaxation will be determined from the time of administration of reversal agent till the the point when TOF ratio is 90-percent.

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Dutta, MD,PGDHR, Study Chair — Sir Ganga Ram Hospital; Subhash Gupta, MD, Study Director — Sir Ganga Ram Hospital; Savitar Malhotra, MD, Principal Investigator — Sir Ganga Ram Hospital
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No